CLINICAL TRIAL: NCT06232564
Title: PELICAN: a Phase II Study of Etoposide-carboplatin Chemotherapy in Combination With Pembrolizumab and Lenvatinib Maintenance in Advanced High-grade Neuroendocrine Tumours (HG-NETs)
Brief Title: A Study of Etoposide-carboplatin in Combination With Pembrolizumab and Lenvatinib Maintenance in HG-NETs
Acronym: PELICAN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1004397
Record Dates: First submitted 2023-12-14; First posted 2024-01-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Neuroendocrine Tumors
Keywords: HG-NETs
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — pembrolizumab; Carboplatin

STUDY DESIGN:
Intervention Model Description: Open Label, Single Arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label, Single Arm, Phase II Study (Experimental): This is an open label, single arm, phase II multicentre study designed to evaluate the efficacy and safety of pembrolizumab in combination with carboplatin and etoposide chemotherapy followed by pembrolizumab and lenvatinib maintenance therapy in patients with HG-NETs who are chemotherapy-naïve for their metastatic disease. The study will be conducted in up to 10 sites and will recruit up to a maximum of 20 evaluable participants.
  Interventions: Combination Product: Pembrolizumab in combination with carboplatin and etoposide chemotherapy followed by pembrolizumab and lenvatinib maintenance therapy

INTERVENTIONS:
Combination Product: Pembrolizumab in combination with carboplatin and etoposide chemotherapy followed by pembrolizumab and lenvatinib maintenance therapy — Pembrolizumab in combination with carboplatin and etoposide chemotherapy followed by pembrolizumab and lenvatinib maintenance therapy

SUMMARY:
This is an open label, single arm, phase II multicentre study designed to evaluate the efficacy and safety of pembrolizumab in combination with carboplatin and etoposide chemotherapy followed by pembrolizumab and lenvatinib maintenance therapy in patients with HG-NETs who are chemotherapy-naïve for their metastatic disease. The study will be conducted in up to 10 sites and will recruit up to a maximum of 20 evaluable participants.

DETAILED DESCRIPTION:
This is an open label, single arm, phase II multicentre study designed to evaluate the efficacy and safety of pembrolizumab in combination with carboplatin and etoposide chemotherapy followed by pembrolizumab and lenvatinib maintenance therapy in patients with HG-NETs who are chemotherapy-naïve for their metastatic disease. The study will be conducted in up to 10 sites and will recruit up to a maximum of 20 evaluable participants.

Patients who satisfy study inclusion criteria will be offered the possibility of participating in the study. A patient information sheet and a written consent form will be offered to every patient. Informed consent must be obtained prior to initiation of any clinical screening procedure that is performed solely for the purpose of determining eligibility for research.

Investigators must ensure that subjects are clearly and fully informed about the purpose of the study, in which they volunteer to participate. In situations where consent cannot be given to subjects, their legally acceptable representatives are clearly and fully informed about the purpose, the subject volunteers to participate. The consent form which will include all elements required by ICH, GCP and applicable regulatory, and will adhere to the ethical principles that have their origin in the Declaration of Helsinki.

Following written content, investigators will assess:

* Patient's Demographics and Medical History;
* Patient's Eligibility Confirmation;

The treatment schedule recognizes an induction phase and a maintenance phase.

Induction Phase. Following informed consent and screening investigations (28 days window) patients will receive 4 cycles of induction chemotherapy with carboplatin (AUC 5mg/ml/min) administered IV alongside etoposide (120 mg/m2) and pembrolizumab (200 mg IV) on day 1 of a 21-days cycle, followed by oral etoposide (100 mg twice daily) on day 2-3 of each cycle.

Maintenance Phase. In patients who achieve a complete, partial response or stable disease following induction, maintenance pembrolizumab (200 mg IV on day 1 every 21 days) and lenvatinib (20 mg PO daily) will start following completion of induction treatment and will continue until unacceptable toxicity, disease progression, withdrawal of consent or completion of 2 years of treatment. In days when Lenvatinib is co-administered with pembrolizumab, lenvatinib should be administered prior to pembrolizumab, ideally in the morning of the study visit. Re-staging by computerised tomography (CT) will be performed 21 days after completion of induction then 9-weekly until study completion. A second, optional tumour biopsy will be taken at C3 Day 1 (+/- 14 days).

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the participant must:

1. Be willing and able to provide written informed consent for the trial.
2. Be 18 years or above of age on day of signing informed consent.
3. ECOG performance status of 0-2.
4. Have histologically or cytologically confirmed diagnosis of poorly differentiated neuroendocrine carcinoma.
5. Have Ki-67 labelling index >20% and/or >20 mitoses/10 high-power fields.
6. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Have had no prior systemic treatment in the metastatic setting.
8. Demonstrate adequate organ function.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Women of childbearing potential must be willing to use a highly effective method of contraception for the course of the study through 120 days after the last dose of Investigational Medicinal Product (IMP).

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Sexually active males must agree to use an adequate method of contraception starting with the first dose of IMP through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

The participant must be excluded from participating in the trial if the participant:

1. Has a diagnosis of large cell and small cell histology of lung origin or Merkel cell carcinoma.
2. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
3. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease and stereotactic radiotherapy to the CNS.
4. Has an active infection requiring systemic therapy.
5. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
6. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA detectable levels) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
7. Has a known history of active Bacillus Tuberculosis (TB).
8. Has a known history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
9. Has a known history of interstitial of lung disease.
10. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Uncontrolled blood pressure (Systolic BP>140 mmHg or diastolic BP >90 mmHg) in spite of an optimized regimen of antihypertensive medication.
13. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug.
14. Bleeding or thrombotic disorders or subjects at risk for severe haemorrhage. The degree of tumour invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe haemorrhage associated with tumour shrinkage/necrosis following lenvatinib therapy.
15. Subjects having >1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
16. Is currently participating and receiving therapy or has participated or is participating in a study of an IMP or used an investigational device within 4 weeks of the first dose of IMP.
17. Has had major surgery within 3 weeks prior to first dose of study treatment.
18. Has a history of hypersensitivity to pembrolizumab, lenvatinib, carboplatin, etoposide or any of their excipients.
19. Has a known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for ≥3 years since initiation of that therapy. (Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.).
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Principal Investigator (PI).
21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through to 120 days after the last dose of IMP.
23. Has received prior therapy with an anti-PD-1, anti-PD-L1 or anti-PD-L2 agent.
24. Has received a live vaccine within 30 days of first dose of IMP administration. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effects of carboplatin, etoposide and pembrolizumab followed by pembrolizumab and lenvantinib maintenance in treatment naïve HG-NETs as measured by RECIST v1.1 criteria. | 2 Years
  To evaluate overall response rates (ORR) as measured by RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Investigation of adverse events from treatment of carboplatin, etoposide and pembrolizumab followed by pembrolizumab and lenvatinib maintenence. | 2 Years
  To evaluate incidence of adverse events of any grade attributable to any of the systemic therapies utilised described according to the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for adverse event reporting. (http://ctep.cancer.gov/reporting/ctc.html).

OTHER OUTCOMES:
To Assess tumour infiltrating lymphocyte profiling | 2 Years
  Assess tumour infiltrating lymphocyte profiling by FACS and clonality assessment by ImmunoSeq.
Immunohistochemistry | 2 Years
  Carry out Multiplex immunohistochemistry for CD8, CD4, FOXP3, PD1, VEGF-A and CD34.
Blood testing for characterisation of cells | 2 Years
  Characterisation of peripheral bloods mononuclear cells for phenotype and clonality.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774